CLINICAL TRIAL: NCT01614925
Title: A Randomized, Controlled, Multicenter Clinical Study Evaluating the Outcomes of Periodontal Surgery in Supra-alveolar-type Defects With or Without Straumann® Emdogain
Brief Title: Safety and Efficacy of Periodontal Surgery in Supra-alveolar-type Defects With or Without Straumann® Emdogain
Status: Terminated | Type: Interventional
Why Stopped: Due to change in strategy and decision not to expand indication.
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR 02/11
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Periodontal Attachment Loss; Periodontal Diseases
MeSH Terms: conditions — Periodontal Attachment Loss; Periodontal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- Emdogain (Experimental): Periodontal surgery with the additional use of Straumann® Emdogain
  Interventions: Device: Emdogain
- Periodontal Surgery (Active Comparator): Periodontal surgery alone
  Interventions: Procedure: Periodontal surgery

INTERVENTIONS:
Device: Emdogain — Periodontal surgery with the additional use of Straumann® Emdogain
  Arms: Emdogain
Procedure: Periodontal surgery — Periodontal surgery alone
  Arms: Periodontal Surgery

SUMMARY:
The primary objective of this study is to demonstrate that in supra-alveolar-type defects (i.e., defects displaying a predominately horizontal pattern of bone loss), periodontal surgery with the additional use of Straumann® Emdogain will result in significantly higher Clinical Attachment Level (CAL) gain compared to periodontal surgery without Straumann® Emdogain.

DETAILED DESCRIPTION:
The following secondary endpoints will be evaluated during the study:

* Change in Gingival Margin (GM) at 12 months after surgery compared to baseline
* Change in Probing Pocket Depth (PPD) at 12 months after surgery compared to baseline
* Comparison of early wound healing index (EHI) at 4 weeks after surgery between treatment groups
* Comparison of post-surgical pain at 4 weeks after surgery between treatment groups
* Change in Bleeding on Probing (BoP) at 12 months after surgery compared to baseline
* Change in root dentin hypersensitivity at 12 months after surgery compared to baseline
* Change in full mouth plaque index (PI) at 12 months after surgery compared to baseline

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have advanced periodontitis:
* presence of supra-alveolar-type defects (i.e., defects displaying a predominantly horizontal pattern of bone loss) at a minimum of two adjacent teeth and a maximum of 7 adjacent teeth (FDI positions 17-27 or 37-47) in either the maxilla or the mandible with a PPD of ≥6 mm at a minimum on one site of the examined teeth
* Teeth must have < Class II mobility
* Teeth must have horizontal bone loss with an intrabony component of <2 mm as defined by radiographic evaluation
* Subjects must have adequate oral hygiene (full mouth plaque index (PI) of <25% at baseline (i.e., following initial non-surgical periodontal therapy)
* Subjects must have adequate control of inflammation (full mouth bleeding on probing (FMBP) of <25% at baseline (i.e., following initial non-surgical periodontal therapy)
* Subjects must have voluntarily signed the informed consent form before any study related procedures
* Subjects must be males and females of at least 18 years of age
* Subjects must be committed to the study and the required follow-up visits
* Subjects must be in good general health as assessed by the investigator at time of surgery

Exclusion Criteria:

Pre-surgical exclusion criteria:

* Subjects with any contraindications for oral surgical procedures
* Subjects with uncontrolled diabetes or other uncontrolled systemic diseases
* Subjects with disorders or treatments that compromise wound healing
* Subjects with medical conditions requiring chronic high dose steroid therapy
* Subjects with bone metabolic diseases
* Subjects with radiation or other immuno-oppressive therapy
* Subjects with infections or vascular impairment at the surgical site
* Subjects who are on antibiotic treatment or chronic anti-inflammatory treatment (≥3 times per week) within 4 weeks prior to surgery.
* Subjects with the presence of oral lesions (such as ulceration, malignancy)
* Subjects with mucosal diseases (e.g., lichen planus, mouth ulcer)
* Subjects with a history of malignant disease in the oral cavity or previous radiotherapy to the head or neck
* Subjects with inadequate oral hygiene or unmotivated for adequate home care
* Subjects that have been treated with an investigational drug or device within the 30 day period immediately prior to surgery on study day 0.
* Subjects who currently smoke
* Female subjects who are nursing, pregnant, or plan to become pregnant

Secondary exclusion criteria:

* Subjects with an osseous defect with an intrabony component of ≥2 mm or involving furcation involvement ≥ class II at the tooth of interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was terminated prematurely.
Period: Overall Study
Arm/Group | Emdogain | Periodontal Surgery
Started | 18 | 17
Completed | 14 | 15
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emdogain | Periodontal Surgery | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (14.0) | 53.9 (13.2) | 52.4 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 14 | 22
  Male | 10 | 3 | 13
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12
  Switzerland | 3 | 3 | 6
  Germany | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Clinical Attachment Level
Description: The change in Clinical Attachment Level (CAL) from Baseline to 12 Months. CAL measurements will be derived from the Probing Pocket Depth (PPD) and Gingival Margin (GM) measurements as follows: CAL = PPD - GM.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Emdogain | Periodontal Surgery
Number analyzed (Participants) | 14 | 15
mm | -2.91 (1.3) | -2.08 (1.32)

2. Secondary Outcome: Change in Gingival Margin (GM) From Baseline to 12 Months
Description: GM was measured by recording the distance from the Cemento-Enamel Junction (CEJ) to the margin of the gingiva at 6 sites (mesio-vestibular, mid-vestibular, disto-vestibular, mesio-oral, mid-oral, disto-oral) on the study teeth. Negative value for GM indicates gingival recession. A positive value for the GM indicates the gingiva was covering the CEJ.
Time Frame: 12 months after baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Emdogain | Periodontal Surgery
Number analyzed (Participants) | 14 | 15
mm | -0.36 (0.84) | -0.27 (1.53)

3. Secondary Outcome: Change in Probing Pocket Depth (PPD) From Baseline to 12 Months
Description: PPD was measured before the area is anaesthetized by recording the distance from the gingival margin to the bottom of the probable pocket at 6 sites (mesio-vestibular, mid-vestibular, disto-vestibular, mesiooral, mid-oral, and disto-oral) on the study teeth.Negative value for PPD indicates reduction of pocket depth.
Time Frame: 12 months after baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Emdogain | Periodontal Surgery
Number analyzed (Participants) | 14 | 15
mm | -2.93 (1.44) | -2.47 (1.12)

4. Secondary Outcome: Early Wound Healing Index (EHI) Assessment at 4 Weeks After Baseline
Description: Postoperative wound healing was assessed by the EHI according to Wachtel et al. [2003] by visual assessment:
  1. complete flap closure - no fibrin line in the interproximal area
  2. complete flap closure - fine fibrin line in the interproximal area
  3. complete flap closure - fibrin clot in the interproximal area
  4. incomplete flap closure - partial necrosis of the interproximal tissue
  5. incomplete flap closure - complete necrosis of the interproximal tissue The outcome measure was the percentage of EHI category 1 (complete flap closure - no fibrin line in the interproximal area)
Time Frame: 4 weeks after baseline
Measure: Number; unit: percentage of EHI category 1
Arm/Group | Emdogain | Periodontal Surgery
Number analyzed (Participants) | 14 | 15
percentage of EHI category 1 | 93 | 100

5. Secondary Outcome: Comparison of Post-surgical Pain at 4 Weeks After Baseline
Description: Visual Analog Scale (VAS) for post-surgical pain, minimum value=0, maximum value=10, higher score means worse outcome
Time Frame: 4 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emdogain | Periodontal Surgery
Number analyzed (Participants) | 14 | 15
score on a scale | 3.21 (9.39) | 3.47 (7.77)

6. Secondary Outcome: Change in Bleeding on Probing (BoP) From Baseline to 12 Months
Description: The presence of BoP was recorded as a binary response on 6 sites (mesio-vestibular, midvestibular, disto-vestibular, mesio-oral, mid-oral, and disto-oral) on the study teeth. The percentage of positive events per total probing sites was calculated for each group. The outcome measure was the change between baseline and 12 months. Negative values indicate a decrease in BoP.
Time Frame: 12 months after baseline
Measure: Number; unit: percentage of BoP change
Arm/Group | Emdogain | Periodontal Surgery
Number analyzed (Participants) | 14 | 15
percentage of BoP change | -36 | -13

7. Secondary Outcome: Change in Root Dentin Hypersensitivity (RDH) From Baseline to 12 Months
Description: RDH was examined by physical testing using cold air as a stimulus. The percentage of positive events per total testing sites was calculated for each group. The outcome measure was the change between baseline and 12 months. Negative values indicate a decrease in RDH.
Time Frame: 12 months after baseline
Measure: Number; unit: percentage of RDH change
Arm/Group | Emdogain | Periodontal Surgery
Number analyzed (Participants) | 14 | 15
percentage of RDH change | -21.4 | -26.7

8. Secondary Outcome: Change in Plaque Index (PI) From Baseline to 12 Months
Description: The PI was recorded according to O'Leary et al. [1972] as a binary response at the mesial, distal, facial and lingual surfaces on the study teeth. The percentage of positive events per total sites was calculated for each group. The outcome measure was the change between baseline and 12 months. Negative values indicate a decrease in PI.
Time Frame: 12 months after baseline
Measure: Number; unit: percentage of PI change
Arm/Group | Emdogain | Periodontal Surgery
Number analyzed (Participants) | 14 | 15
percentage of PI change | 14.7 | 13.4

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Emdogain | Periodontal Surgery
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 1/18 | 1/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emdogain (N=18) | Periodontal Surgery (N=17)
Tooth hypersensitivity (General disorders) | 0 (0) | 1 (1)
Aphthous ulcer (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. This sponsor decision was based on commercial reasons and not linked to any safety concerns or new scientific knowledge.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No